CLINICAL TRIAL: NCT07036133
Title: A Phase 1, Open-Label, Multicenter Study to Evaluate the Pharmacokinetics and Safety of Pralatrexate in Patients With Advanced Solid Tumor or Hematological Malignancy and Either Normal Hepatic Function or Mild, Moderate, or Severe Hepatic Impairment
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of Pralatrexate in Patients With Advanced Solid Tumor or Hematological Malignancy and Either Normal Hepatic Function or Mild, Moderate, or Severe Hepatic Impairment
Acronym: SPI-FOL-102
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOL-102
Record Dates: First submitted 2025-03-18; First posted 2025-06-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors; Hematologic Malignancies
Keywords: Pralatrexate
MeSH Terms: conditions — Hematologic Neoplasms | interventions — 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label treatment with Pralatrexate (Other): Pralatrexate will be administered based on Child-Pugh Classification of liver impairment.
  Interventions: Drug: Pralatrexate Injection

INTERVENTIONS:
Drug: Pralatrexate Injection — Pralatrexate will be administered based on Child-Pugh Classification of liver impairment

SUMMARY:
This purpose of this study is to help to evaluate the pharmacokinetic (PK) profile of pralatrexate when administered to patients with various degrees of hepatic impairment and to evaluate the safety and establish the dosing recommendations for pralatrexate administered once weekly for 6 weeks of every 7-week treatment cycle in patients with hepatic impairment. Pharmacokinetics (or PK) is the study of how your body absorbs, breaks down, and removes a study drug.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center study to evaluate the PK and safety of pralatrexate in patients with advanced solid tumor or hematological malignancy with normal hepatic function or mild, moderate, or severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be willing and capable of giving written Informed Consent and must be able to adhere to dosing and visit schedules as well as meet all study requirements
* Patient is diagnosed with advanced solid tumor or hematological malignancy.
* Patient is at least 18 years of age and has a life expectancy of at least 6 months.
* Patient has normal or abnormal hepatic function as defined by normal, mild (Child-Pugh A), moderate (Child-Pugh B ), or severe (Child-Pugh C) liver impairment
* Patient has adequate hematologic and renal function as defined by:

Absolute neutrophil count (ANC) ≥1000/μL Platelet count ≥100,000/μL Creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥50 mL/min

* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patient is willing to practice 2 forms of contraception, one of which must be a barrier method, from study entry until at least 30 days after the last dose of pralatrexate
* Females of childbearing potential must have a negative pregnancy test within 30 days prior to enrollment. Females who are postmenopausal for at least 1 year (defined as more than 12 months since last menses) or who are surgically sterilized do not require this test.

Exclusion Criteria:

* Patient has had previous exposure to pralatrexate
* Patient has used any investigational drugs, biologics, or devices within 30 days prior to study treatment or plans to use any of these during the course of the study.
* Patient has an active, uncontrolled infection, underlying medical condition, or other serious illness that would impair the patient's ability to receive the protocol-defined treatment.
* Patient has known or suspected intolerance or hypersensitivity to the investigational product or any related compound.
* Patient has congestive heart failure at Class III/IV according to the New York Heart Association (NYHA) Functional Classification
* Patient has had major surgery within 30 days prior to enrollment.
* Patient with central nervous system (CNS) metastases
* Patient is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic (PK) profile of pralatrexate. | During week 1 of the first cycle of treatment (each cycle is 7 weeks).
  Blood will be collected to evaluate the pharmacokinetic (PK) profile of pralatrexate (plasma concentration levels) when administered to patients with various degrees of hepatic impairment.

SECONDARY OUTCOMES:
To evaluate the safety of pralatrexate | This will be evaluated during the study through 14(±3) days after the last dose in Cycle 1, or 35(±5) days after the final dose in any cycle or until all treatment-related AEs have resolved or returned to Baseline/Grade
  The number and severity of treatment-related adverse events. This will be as assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) scale, Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Erard Gilles, MD, MSc, Study Director
Locations (4):
- United States (4):
  - TOI Clinical Research, Cerritos, California
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Gabrail Cancer Center, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No